# A Study Protocol for a Randomised Controlled Trial Evaluating the Benefits from Bimodal Solution with Cochlear Implant and Hearing Aid vs. Bilateral Hearing Aids in Patients with Asymmetric Speech Identification Scores.

Trial Registration Number: NCT04919928 (ClinicalTrials.gov)

Updated: 21.08.22

# A Study Protocol for a Randomised Controlled Trial Evaluating the Benefits from Bimodal Solution with Cochlear Implant and Hearing Aid vs. Bilateral Hearing Aids in Patients with Asymmetric Speech Identification Scores.

Yeliz Jakobsen<sup>1,2\*</sup>, Lou-Ann Christensen Andersen<sup>3</sup>, Jesper Hvass Schmidt<sup>1,2</sup>

#### Affiliation

- <sup>1</sup> Research Unit for ORL Head & Neck Surgery and Audiology, Odense University Hospital, Odense, Denmark; University of Southern Denmark, Odense, Denmark
- <sup>2</sup> OPEN, Odense Patient data Explorative Network, Odense University Hospital, Odense, Denmark.
- <sup>3</sup>Department of Ophthalmology, Lillebaelt Hospital, Vejle Hospital.
- \*Correspondence to Dr. Yeliz Jakobsen; Yeliz.jakobsen@rsyd.dk

Date: Sunday, 21st August 2022

Version: 3

#### **Abstract**

#### Introduction

Cochlear implant (CI) and hearing aid (HA) in a bimodal solution (CI + HA) is compared to bilateral HAs (HA +HA) to test if the bimodal solution result in better speech intelligibility and self-reported quality of life.

## Methods and Analysis

This randomised controlled trial (RCT) is conducted in Odense University Hospital,
Denmark. Sixty adult bilateral HA users referred for CI surgery is enrolled if eligible and
undergo: audiometry, speech perception in noise (HINT: Hearing in Noise Test), Speech
Identification Scores (SIS) and video head impulse test (v-HIT). All participants will receive
new replacement HAs. After one month they will be randomly assigned (1:1) to the
intervention group (CI+HA) or to the delayed intervention control group (HA+HA). The
intervention group (CI+HA) will receive a CI on the ear with a poorer speech recognition

score and continue using the HA on the other ear. The control group (HA+HA) will receive

a CI after a total of 4 months of bilateral HA use.

The primary outcome measures are Speech intelligibility measured objectively with HINT

(sentences in noise) and DANTALE I (words) and subjectively with the Speech, Spatial

and Qualities of Hearing scale questionnaire (SSQ-12). Secondary outcomes are patient

reported Health-Related Quality of Life (HRQoL) scores assessed with the Nijmegen

Cochlear Implant Questionnaire (NCIQ), the Tinnitus Handicap Inventory (THI) and

Dizziness Handicap Inventory (DHI). Third outcome is listening effort assessed with pupil

dilation during HINT

In conclusion, the purpose is to improve clinical decision-making for CI candidacy and

optimize bimodal solutions.

**Ethics and Dissemination** 

This study protocol was approved by the Ethics Committee Southern Denmark project ID

S-20200074G. All participants are required to sign an informed consent form.

This study will be published upon completion in a peer-reviewed publications and scientific

conferences.

Trial Registration Number: NCT04919928 (ClinicalTrials.gov)

3

## Strengths and Limitations of This Study

- The study uses comprehensive measures of self-reported outcomes as well as objective tests of speech intelligibility.
- Listening effort controlled with pupillometry during objective tests of speech intelligibility.
- Open label RCT (blinding is not possible due to visibility of the CI).
- Possible large drop rates if new HAs improve speech intelligibility to an extent that
   CI treatment is rejected or postponed.

## Introduction

## Background

Cochlear implants (CIs) have been used to restore hearing in individuals with severe to profound sensorineural hearing loss. Initially, most patients receiving a cochlear implant were profoundly deaf in both ears. (1, 2) However, recently it has become more common to implant patients with significant residual hearing in the affected ear, as well as in patients with asymmetric hearing loss and single-sided deafness, with significant residual hearing or normal hearing on the contralateral side.(3, 4) A CI in one ear and a HA in the other ear can provide enhanced hearing performance in patients with asymmetrical hearing.(5, 6) The combination of CI and HA is referred to as bimodal hearing or bimodal solution.(7)

# CI Candidacy

In the UK, The National Institute for Health and Care Excellence (NICE) have listed guidelines for cochlear implantation and recommends that unilateral CI is offered to patients

with severe to profound deafness who do not receive adequate benefit from acoustic hearing aids. Severe to profound deafness is defined as pure-tone audiometric threshold  $\geq$  80 dB HL at 2 or more frequencies (500 Hz, 1,000 Hz, 2,000 Hz, 3,000 Hz and 4,000 Hz). Another criteria is that SIS< 50% in the ear considered for implantation and in best aided condition SIS $\leq$ 60%(8).

The Danish CI candidacy criteria consists of SIS (without HAs, measured with headphones) ≤45% and a SIS ≤65% (in best aided condition) in the ear considered for implantation using DANTALE I monosyllabic word-lists.(9) Additional testing to evaluate speech understanding is assessed by HINT.(10, 11)

The recommendation for a CI might be less clear for patients with asymmetric hearing because they may not fall into the traditional referral criteria but would likely benefit from a CI. It is therefore necessary to establish more evidence to support the effectiveness of bimodal CI+HA versus HAs in patients with asymmetric hearing.

## Bimodal Solution vs. Bilateral HAs

Normal hearing listeners (NH) benefit from listening with two ears, which help them understand speech in noise and identify sound location.

Benefits from listening with two ears include: head shadow effect, binaural summation, binaural squelch, localization and spatial release from masking.(12-15)

Patients with hearing loss often do not have these benefits, and they are often not accessible to CI patients. (15)Many bimodal CI and HA users are missing these benefits because the devices are unsynchronized.(16)

Until now it is unknown when to introduce the bimodal solution and making sure that patients are well-fitted with hearing aids when they are given the candidacy assessment.

The question is if the bimodal benefits are bigger than the bilateral hearing aid condition when they are well fitted?

This study will therefore support and strengthen the preoperative clinical decision to recommend a bimodal solution with a CI and a HA versus the continuous use of bilateral HAs. This may offer the patient faster and more effective treatment because delaying the surgery may not be beneficial.

## Patient-Reported Outcome Measures

Benefits of the CI are measured subjectively with Patient-Reported Outcome Measures (PROMs) as SSQ12, NCIQ, THI and DHI.(17-24)

The validity and reproducibility of the Danish version of THI has been reported(24). SSQ12, DHI, NCIQ have all been translated into Danish and backward translated to English following a cultural adaption and pilot-testing to ensure correct understanding of the questionnaires. Test-retest reliability has been assessed as well.(18, 20, 22)

# Listening Effort

Patients with CI often experience high levels of listening effort, they often report that understanding speech causes high levels of increased sustained effort which results in feelings of fatigue.(25) These feelings may lead patients to withdraw socially due to the stresses involved in communication even though they may not specifically report difficulties with speech understanding.(19)

Effort in listeners with NH can be reflected by the relationship between speech intelligibility and pupil-dilation.(26) Listening effort has been defined as the "Deliberate allocation of

mental resources to overcome obstacles in goal pursuit when carrying out a task" and is the basis for the Framework for Understanding Effortful Listening (FUEL) model.(27) Understanding speech in challenging hearing environments results in increased auditory and cognitive processing which can be observed objectively by measuring the pupil dilation during speech perception in noise, in a task such as the HINT(28-30)

# **Rationale and Objectives**

This randomised controlled trial is designed to improve clinical decision-making for CI candidacy for patients with asymmetric hearing. It is necessary to establish more evidence to support the effectiveness and the fitting optimization of bimodal CI+HA versus HAs in patients with asymmetric hearing.

The first objective of the study is to evaluate the subjective (SSQ12) and objective (Hearing In Noise Test (HINT) which is word and sentence based and DANTALE I, which is monosyllabic word-based) benefits of a bimodal solution (CI+HA) compared to (HA+HA).

The second objective is to compare and evaluate patient self-reported outcomes with NCIQ, THI and DHI in the intervention group (CI+HA) with the control group (HA+HA). The third objective is to evaluate if listening effort, hypothesized to cause fatigue, can be measured objectively by HINT with pupillometry.

To minimize listening effort and optimize the fitting of bimodal solution the CI fitting and loudness balancing on individual level will be evaluated.(2, 31, 32)

# **Methods and Analysis**

## Study Design, Ethics and Registration

This study is a prospective randomised controlled trial based on a single centre conducted in Odense University Hospital, Denmark. The study started 01/02/2022 and is expected to end 30/07/2024. It was successfully registered at ClinicalTrials.gov with registration number: NCT04919928.

This study has been approved at Research Ethics Committee Southern Denmark (Projekt-ID: S-20200074G) 21<sup>st</sup> August 2020 to 31<sup>st</sup> December 2024.

## Study Population

Sixty participants with bilateral hearing-loss and asymmetric speech identification scores referred for CI surgery will be included (Figure 1).

## **Inclusion Criteria**

- Adults >18 years old.
- Fluent in Danish, including reading and writing
- Acquired post-lingual deafness
- Use of bilateral HAs for at least one year prior to evaluation for cochlear implantation candidacy. This to ensure, that both ears have received auditive stimulation
- PTA > 40 dB HL in the ear considered for CI implantation and PTA≥40 and ≤ 70dB
   HL in the contralateral ear in best aided condition, in quiet and in noise and in free field.

SIS <70% in best aided condition in the ear considered for CI implantation and SIS</li>
 ≥30% and ≤70% in best aided condition in the contralateral ear, in quiet and in noise and in free field.

#### **Exclusion Criteria**

- Vestibular loss in the ear not considered for CI implantation
- Surgical issues interfering with the site of implantation or anatomical contraindications such as cochlear malformations, which will be determined using MRI or CT-scans.
- Auditory nerve lesions.
- Central auditory pathway pathologies.
- Otosclerosis.
- Single sided deafness (SSD).

## Setup

A timeline of the study is shown in (Figure 2).

All enrolled participants will be tested with audiometry and v-HIT to determine hearing thresholds and status of balance function during the first visit. Patients will receive new replacement HAs. These HAs will be fitted during the second visit and if necessary refitted at every visit in the clinic throughout the study. The baseline measurements will be conducted when both groups have used the new replacement HAs to ensure acclimatisation. The measurements are SIS in quiet and in noise with a signal-to-noise ratio (SNR) of 0dB using DANTALE I speech material. The speech and masking white noise

stimulus will be presented at 65 dB SPL in the free field. Stimuli will be presented as auditory stimuli only as well as with visual cues, the latter to allow participants to use lipreading cues. Pupillometry variables are Peak Pupil Dilation (PPD), Mean Pupil Dilation (MPD), peak-time and standard deviation using HINT (sentences and words).

The HINT sentences are presented at a speech level of 65dB and initially an adaptive SNR is used to identify the SNR of 70% correct word recognition. The SNR at 70% correct word recognition is used as a fixed SNR during HINT test. The noise is multi-talker babble noise, in free field, tested in best aided condition. The pupillometry glasses is the Oticon Medical Pupil Labs glasses.

## Recruitment, Stratification, Randomisation and Allocation

All eligible participants will sign a written, informed consent in clinic after receiving verbal and written study information in Danish. The Danish consent form is available online at the Odense University Hospital Research Unit website.(33)

To ensure acclimatisation, participants will receive new replacement HAs fitted with the National Acoustic Laboratories (NAL) -non-linear (NL)2 fitting algorithm one month before the experiment.

They will then undergo stratification, depending on the hearing thresholds. One group will consist of participants with PTA  $\geq$  70dB HL; and the other group will consist of subjects with PTA  $\leq$  70dB HL and  $\geq$  40 dB HL according to the inclusion criteria. The reason for this stratification is because pre-operative hearing thresholds may affect the measured outcomes in the study. Stratification ensures that both the intervention group and the control group will have an equal distribution of patients with profound hearing loss on the ear considered for implantation.

Then the participants will be randomly allocated into two groups: the intervention group (CI+HA) and the control group (HA+HA) according to 1:1 ratio using a blocked randomisation with randomly varying block size (4 or 6).

This randomisation will be accomplished using a computer-generated random sequence in Research Electronic Data Capture (REDCap), hosted by Odense Patient Explorative Network (OPEN) in the Region of Southern Denmark and developed by Vanderbilt University, Nashville, Tennessee, United States.(34)

REDCap will also be used to send out the questionnaires to the participants' online mailbox (called Eboks in Denmark) throughout the study (see timeline (Figure 2)) and automatically save the data.

Participants will have the opportunity to return to their original HAs if they prefer to do so after one-month of acclimatisation.

## **Control Group**

Thirty patients, who will be age-matched, randomised and allocated to the control group HA+HA will continue the use of the new replacement HAs for another three months (total four months of new replacement HA+HA use), serving as the delayed intervention control group.

# Intervention Group

Thirty patients, who will be age-matched, randomised and allocated to the intervention group CI+HA will undergo surgery as soon as possible after the HA acclimatisation period.

## **HA** Fitting

The participant will receive either Phonak (Phonak Link M) or GN (ReSound LiNX Quattro or Resound ENZO Q) based on their personal preference. Both these HA models can be fitted with a CI by Advanced Bionics and Cochlear, respectively.

The HAs will be fitted according to NAL-NL2 procedures prescriptive fitting formula, which optimizes audibility in the bimodal solution(2) and will be verified with REM (Real Ear Measurement) to ensure that the HA is providing adequate gain and then further adjusted for comfort based on patient feedback.(35)

The new HAs will be prescribed to the patients free of charge and future service will also be free of charge.

Participants can drop out of the study if they do not want CI surgery. Collected data will be analysed if the patient still consents.

# CI fitting

The CI will be selected depending on the participant's HA selection; that is, the CI that is compatible with the HA will be selected in order to ensure the most optimal bimodal fitting. One-month post-surgery, the CI will be activated according to the settings and stimulation strategy based on patient's feedback. The CI will then be fitted with the HA according to the bimodal fitting formula allowing the HA to keep the NAL-NL2 fitting along with the wireless connection with the CI. (36, 37)

Patients hearing thresholds will be tested on CI activation day. The residual hearing will not be stimulated in this study.

All participants are offered standard rehabilitation with a speech therapist, including three visits a week up to 10 weeks following the initial fitting.

The training focuses on learning to identify different sounds from the environment and word discrimination.

The new CI will also be prescribed to the patients free of charge and future service will be free of charge as well.

## Loudness Balancing

At 3- months follow-up the post-surgery complications will be evaluated and the levels in the CI will be adjusted if necessary.

In the loudness balancing procedure, the patient will have both the hearing aid and CI activated and at the 6-month follow-up, when the CI mapping levels are stable, patients will be randomised and assigned to one of three bimodal fitting groups:

Group A) will not complete any specific loudness balancing procedures, CI and HA will be fitted based on individual feedback from the patient.

Group B) will be fitted/finetuned using a bimodal loudness balancing task at a medium input level and adjusted based on the patient feedback. The audiologist will present a midlevel sound (approx. 55dB SPL (sound pressure level)) at the center-speaker.

Group C) will be fitted/finetuned using a bimodal loudness balancing task as group B but the audiologist will play three levels and adjust the gain for three input levels (soft, medium, and loud) according to the patient feedback.

For both groups B and C, the patient will be given a 'Bimodal Fusion' illustration (see Figure 3) and asked to provide feedback about the location of the sound by tracing over the line of

the head. The HA gain will be adjusted using the bimodal adjustment option until the patient reports that the sounds are perceived at the center of the head.(24)

## **Primary Outcome**

Primary outcomes are Speech intelligibility scores measured objectively with HINT (sentences and words) and DANTALE I and subjectively with Speech, Spatial and Qualities of Hearing scale (SSQ-12). (9, 10, 22)

## Secondary Outcome

Patient reported outcomes scores assessed with the Nijmegen Cochlear Implant

Questionnaire (NCIQ), The Tinnitus Handicap Inventory (THI) and Dizziness Handicap

Inventory (DHI). (18, 20, 24)

## Third Outcome

Listening effort assessed with pupil dilation with HINT.(10)

## **Statistics**

## Power calculation

Power calculations with a power of 0.8 with a significance level of 0.05 have been made with STATA IC-15 using standard deviations for the HINT test and expected effect size (38) the NCIQ(18), and the SSQ (internal communication with BEAR (Better Hearing Rehabilitation) study on hearing aid use in Denmark) (Table 1). An estimated within participant standard deviation from the BEAR study of 1,9 in an HA population using the

SSQ-12 is used to calculate the sample size. A difference of 1,4 will require 30 participants in each arm. The effect size is expected to be larger in the CI group which will lower the number of required subjects even further.

Based on this, 30 participants must be enrolled in each arm. Additional six patients (20%) in each arm will be enrolled in the study to account for dropouts.

| Test | SD pre | SD post | Expected difference between the two treatment arms | Minimum<br>required group<br>size |
|---|---|---|---|---|
| 1. HINT | 6.3% | 6.3% | 5% | 26 |
| 2. NCIQ - basic sound perception | 14.4 | 23.5 | 53 | 4 |
| 2. NCIQ | 13.4 | 19.6 | 34 | 6 |
| 2. NCIQ - speech perception | 18.8 | 17.8 | 17 | 20 |
| 2.NCIQ Self-esteem | 20.1 | 16.4 | 22 | 13 |
| 2.NCIQ Activity | 23.0 | 15.9 | 27 | 10 |
| 2.NCIQ Social Interactions | 19.8 | 14.5 | 25 | 9 |
| 3. SSQ Total | 1.9 | 1.9 | 1.4 | 30 |

Table 1: Power calculations for the desired tests. Estimated within participant standard deviations (SD pre and SD post) with expected difference and the calculated required group size.

# **Definition of Analysis Sets**

Strategy for intention to treat analysis with incomplete observations.(39)

- Attempt to follow-up on all randomised participants, even if they withdraw from allocated treatment.
- 2. Perform a main analysis of all observed data that are valid under a plausible assumption about the missing data.
- 3. Perform sensitivity analyses to explore the effect of deviations from the assumption made in the main analysis.
- 4. Account for all randomised participants, at least in the sensitivity analyses.

## Analysis specification

A constrained linear mixed model is used to analyse the outcome.

The model will include randomisation group (CI+HA / HA+HA) and time (baseline/follow-up) and their interaction as fixed effects along with the threshold strata that were used in stratifying the randomisation. The model is constrained so that the mean at baseline agrees across the two treatment groups adjusted for threshold stratum, which is reasonable due to the randomisation of implant fitting. Patient ID will be included as a random effect to account for the repeated measurements.

Secondary outcomes will be analysed analogously in a constrained linear mixed model adjusting for randomisation strata. Model validation checks will be undertaken as described above, switching to bootstrapping the standard errors when model assumptions are rejected.

Covariates such as age and gender will be included in all models.

## Sensitivity analysis

Inclusion is performed conditional on Pure Tone Average (PTA) (from 0.5 to 4 kHz) PTA > 40 dB HL and SIS <50% in the ear considered for CI implantation and <70% in the best-aided condition which may lead to a truncation effect in the distribution of baseline measurements. To address this, an analysis of covariance (ANCOVA) model conditioning on the baseline will be used to obtain a sensitivity analysis estimate for the main outcome.(40)

The statistical analysis plan is attached as "supplementary file" along with the Data Description listed in Appendix A.

#### **Patient and Public Involvement**

A focus-group interview was established with six cochlear implant patients. The patients commented on their decision to transition from HA to CI. Based on the feedback from the focus group, the research questions were developed.

The patients also reported problems with adjustments of the CI, when meeting the audiologist for CI adjustment controls.

#### **Ethics and Dissemination**

Ethics approval for the conduct of this study was obtained from the Ethics Committee Southern Denmark, 21st August 2020 project ID S-20200074G.

The project is approved by the Danish Data Protection Agency (file no. 20/22868) in Region South Denmark.

All participants are treated according to current clinical standards regardless of the randomised study participation. The participants are volunteers and can at any moment withdraw their participation in the study without affecting their current or future treatment rights.

The Informed Consent form will be found online as an online supplementary file and it will be signed by all participants willing to participate the study and stored in their electronic journals in Department of Audiology, Odense University Hospital. All patients are given both oral and written information about the study.

## Results

Results will be presented at national and international congresses and published in the scientific literature for the attention of professional and scientific audiences on behalf of all study sites and collaborators. A lay summary report will be published for patients and members of the public.

#### **Footnotes**

#### **Authors' Contributions:**

YJ and JHS are involved in the conception of the study. LCA and JHS wrote the grant application. LCA and JHS wrote the draft of the manuscript. JHS designed and revised the draft of the methodological content. YJ reviewed and JHS critiqued the manuscript. YJ and JHS approved the final manuscript6

#### Funding:

This study is funded by William Demant Foundation grant no. 19-3470 and Interfond grant no. 33.188

#### **Competing Interests:**

None declared

#### **Contributorship Statement/Acknowledgements:**

We are very thankful of the academic English editing of Ph.D. Kathleen F. Faulkner and Assistant Professor Lindsey Van Yper

We are grateful for the contribution from the patient advisers.

#### **Protocol and Registration:**

This study is registered in ClinicalTrials.gov: NCT04919928

## **Reference List**

1. Morera C, Manrique M, Ramos A, Garcia-Ibanez L, Cavalle L, Huarte A, et al. Advantages of binaural hearing provided through bimodal stimulation via a cochlear implant and a conventional hearing aid: a 6-month comparative study. Acta Otolaryngol. 2005;125(6):596-606.

- 2. Vroegop JL, Goedegebure A, van der Schroeff MP. How to Optimally Fit a Hearing Aid for Bimodal Cochlear Implant Users: A Systematic Review. Ear Hear. 2018;39(6):1039-45.
- 3. Firszt JB, Holden LK, Reeder RM, Cowdrey L, King S. Cochlear implantation in adults with asymmetric hearing loss. Ear Hear. 2012;33(4):521-33.
- 4. van Zon A, Peters JP, Stegeman I, Smit AL, Grolman W. Cochlear implantation for patients with single-sided deafness or asymmetrical hearing loss: a systematic review of the evidence. Otol Neurotol. 2015;36(2):209-19.
- 5. Thompson NJ, Dillon MT, Buss E, Rooth MA, King ER, Bucker AL, et al. Subjective Benefits of Bimodal Listening in Cochlear Implant Recipients with Asymmetric Hearing Loss. Otolaryngol Head Neck Surg. 2020;162(6):933-41.
- 6. Dillon MT, Buss E, Rooth MA, King ER, McCarthy SA, Bucker AL, et al. Cochlear Implantation in Cases of Asymmetric Hearing Loss: Subjective Benefit, Word Recognition, and Spatial Hearing. Trends Hear. 2020;24:2331216520945524.
- 7. van Loon MC, Smits C, Smit CF, Hensen EF, Merkus P. Cochlear Implantation in Adults With Asymmetric Hearing Loss: Benefits of Bimodal Stimulation. Otol Neurotol. 2017;38(6):e100-e6.
- 8. The National Institute for Health and Care Excellence (NICE) 2019.
- 9. Elberling C, Ludvigsen C, Lyregaard PE. DANTALE: a new Danish speech material. Scand Audiol. 1989;18(3):169-75.
- 10. Nielsen JB, Dau T. The Danish hearing in noise test. Int J Audiol. 2011;50(3):202-8.
- 11. Zhang E, Coelho DH. Beyond Sentence Recognition in Quiet for Older Adults: Implications for Cochlear Implant Candidacy. Otol Neurotol. 2018;39(8):979-86.
- 12. Bronkhorst AW, Plomp R. The effect of head-induced interaural time and level differences on speech intelligibility in noise. J Acoust Soc Am. 1988;83(4):1508-16.
- 13. Bronkhorst AW, Plomp R. Binaural speech intelligibility in noise for hearing-impaired listeners. J Acoust Soc Am. 1989;86(4):1374-83.
- 14. Bronkhorst AW, Plomp R. A clinical test for the assessment of binaural speech perception in noise. Audiology. 1990;29(5):275-85.
- 15. Choi SJ, Lee JB, Bahng J, Lee WK, Park CH, Kim HJ, et al. Effect of low frequency on speech performance with bimodal hearing in bilateral severe hearing loss. Laryngoscope. 2016;126(12):2817-22.
- 16. Balkenhol T, Wallhäusser-Franke E, Rotter N, Servais JJ. Cochlear Implant and Hearing Aid: Objective Measures of Binaural Benefit. Front Neurosci. 2020;14:586119.
- 17. Devlin NJ AJ. Getting the most of proms: putting health outcomes at the heart of NHS decision-making. London, Kings Fund and Office of Health Economics 2010.
- 18. Hinderink JB, Krabbe PF, Van Den Broek P. Development and application of a health-related quality-of-life instrument for adults with cochlear implants: the Nijmegen cochlear implant questionnaire. Otolaryngol Head Neck Surg. 2000;123(6):756-65.
- 19. Hughes SE, Hutchings HA, Rapport FL, McMahon CM, Boisvert I. Social Connectedness and Perceived Listening Effort in Adult Cochlear Implant Users: A Grounded Theory to Establish Content Validity for a New Patient-Reported Outcome Measure. Ear Hear. 2018;39(5):922-34.
- 20. Jacobson GP, Newman CW. The development of the Dizziness Handicap Inventory. Arch Otolaryngol Head Neck Surg. 1990;116(4):424-7.
- 21. Mertens G, De Bodt M, Van de Heyning P. Cochlear implantation as a long-term treatment for ipsilateral incapacitating tinnitus in subjects with unilateral hearing loss up to 10 years. Hear Res. 2016;331:1-6.

- 22. Noble W, Jensen NS, Naylor G, Bhullar N, Akeroyd MA. A short form of the Speech, Spatial and Qualities of Hearing scale suitable for clinical use: the SSQ12. Int J Audiol. 2013;52(6):409-12.
- 23. Servais JJ, Hörmann K, Wallhäusser-Franke E. Unilateral Cochlear Implantation Reduces Tinnitus Loudness in Bimodal Hearing: A Prospective Study. Front Neurol. 2017;8:60.
- 24. Zachariae R, Mirz F, Johansen LV, Andersen SE, Bjerring P, Pedersen CB. Reliability and validity of a Danish adaptation of the Tinnitus Handicap Inventory. Scand Audiol. 2000;29(1):37-43.
- 25. Winn MB, Edwards JR, Litovsky RY. The Impact of Auditory Spectral Resolution on Listening Effort Revealed by Pupil Dilation. Ear Hear. 2015;36(4):e153-65.
- 26. Zekveld AA, Kramer SE, Festen JM. Pupil response as an indication of effortful listening: the influence of sentence intelligibility. Ear Hear. 2010;31(4):480-90.
- 27. Pichora-Fuller MK, Kramer SE, Eckert MA, Edwards B, Hornsby BW, Humes LE, et al. Hearing Impairment and Cognitive Energy: The Framework for Understanding Effortful Listening (FUEL). Ear Hear. 2016;37 Suppl 1:5s-27s.
- 28. Ohlenforst B, Zekveld AA, Lunner T, Wendt D, Naylor G, Wang Y, et al. Impact of stimulus-related factors and hearing impairment on listening effort as indicated by pupil dilation. Hear Res. 2017;351:68-79.
- 29. Wendt D, Koelewijn T, Książek P, Kramer SE, Lunner T. Toward a more comprehensive understanding of the impact of masker type and signal-to-noise ratio on the pupillary response while performing a speech-in-noise test. Hear Res. 2018;369:67-78.
- 30. Eckert MA, Teubner-Rhodes S, Vaden KI, Jr. Is Listening in Noise Worth It? The Neurobiology of Speech Recognition in Challenging Listening Conditions. Ear Hear. 2016;37 Suppl 1(Suppl 1):101s-10s.
- 31. Francart T, McDermott HJ. Psychophysics, fitting, and signal processing for combined hearing aid and cochlear implant stimulation. Ear Hear. 2013;34(6):685-700.
- 32. Wang Y, Naylor G, Kramer SE, Zekveld AA, Wendt D, Ohlenforst B, et al. Relations Between Self-Reported Daily-Life Fatigue, Hearing Status, and Pupil Dilation During a Speech Perception in Noise Task. Ear Hear. 2018;39(3):573-82.
- 33. Jakobsen Y, Schmidt JH. Behandling af nedsat hørelse med cochlear implantat (CI) og høreapparat i kombination i forhold til høreapparater alene. 2022.
- https://ouh.dk/media/vwihy4wi/deltagerinformation-for-bimodal-medlodtr%C3%A6kning.pdf (accessed 21. Aug. 2022).
- 34. Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009;42(2):377-81.
- 35. Digeser FM, Engler M, Hoppe U. Comparison of bimodal benefit for the use of DSL v5.0 and NAL-NL2 in cochlear implant listeners. Int J Audiol. 2020;59(5):383-91.
- 36. Cuda D, Murri A, Mainardi A, Chalupper J. Effectiveness and efficiency of a dedicated bimodal fitting formula. Audiol Res. 2019;9(1):219.
- 37. Stronks HC, Briaire JJ, Frijns JHM. The Temporal Fine Structure of Background Noise Determines the Benefit of Bimodal Hearing for Recognizing Speech. J Assoc Res Otolaryngol. 2020;21(6):527-44.
- 38. Poissant SF, Bero EM, Busekroos L, Shao W. Determining cochlear implant users' true noise tolerance: use of speech reception threshold in noise testing. Otol Neurotol. 2014;35(3):414-20.

- 39. White IR, Horton NJ, Carpenter J, Pocock SJ. Strategy for intention to treat analysis in randomised trials with missing outcome data. Bmj. 2011;342:d40.
- 40. Liu GF, Lu K, Mogg R, Mallick M, Mehrotra DV. Should baseline be a covariate or dependent variable in analyses of change from baseline in clinical trials? Stat Med. 2009;28(20):2509-30.